CLINICAL TRIAL: NCT01404247
Title: Spectral Domain Optical Coherence Tomography Imaging of the Eyes of Neonates
Acronym: OCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Sherwin Isenberg, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 14069-01
Record Dates: First submitted 2011-05-10; First posted 2011-07-28 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Retinal Diseases; Optic Nerve Diseases
Keywords: retina; optic nerve; fovea; Eyes; Neonates
MeSH Terms: conditions — Retinal Diseases; Optic Nerve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OCT imaging in neonates (Experimental): OCT imaging of all neonates, 38-42 weeks, enrolled in this study
  Interventions: Other: Observational: to better characterize the retina and optic nerve in newborns using spectral domain optical coherence tomography (s-oct).; Procedure: OCT imaging.

INTERVENTIONS:
Other: Observational: to better characterize the retina and optic nerve in newborns using spectral domain optical coherence tomography (s-oct). — The OCT technician will attempt to image the eyes of neonates. The neonate may be given Cyclomydril ophthalmic solution, if needed for dilation. Cyclomydril dosing for this study is 1 drop every 5 minutes times 2.
Procedure: OCT imaging. — All newborns meeting eligibility requirements will undergo spectral domain optical coherence tomography imaging in order to better characterize the retina and optic nerve in newborns
  Other Names: OCT imaging

SUMMARY:
Brief Summary

The purpose of this study is to better characterize the retina and optic nerve in newborns using spectral domain optical coherence tomography (s-oct). This new technology provides a very detailed cross-section picture of the cellular layers in the retina and a 3-dimensional picture of the optic nerve head and the fovea (the center of the retina that provides the most accurate vision). These images have been used by doctors for more than 5 years to help diagnose and treat adults with eye diseases, such as macular degeneration, diabetic retinopathy, retinal detachments, and melanoma. But, it has never been studied in newborns. In newborns, it would potentially help in the diagnoses of glaucoma, optic nerve hypoplasia, foveal hypoplasia, and colobomata among many other disorders. Prior to diagnosing disorders, it is necessary to establish normal values. It is the purpose of this investigation to study the retina and optic nerves in neonates to establish normal values.

After a parent of a normal newborn provides a written consent, the baby will be taken to the Eye Clinic where the instrument is located. The baby will be swaddled in one or more blankets as needed. The infants will be held in front of the instrument by a nurse. The technician will move the lens of the instrument to about 2 to 4 inches from the baby's eye. The mild light from the instrument will then enter the eye for a few seconds to obtain the desired image. The image can be captured through an immobile eye within 5 seconds. If the baby is fussy, he or she may be given a few drops of a sugar (sucrose) solution on a pacifier for calming. Although the images can usually be secured through a normal pupil, if the pupil is found to be too small, two drops of Cyclomydril will be placed on the eye for dilation. This is the eye drop used everyday in the Eye Clinic and nursery to dilate the pupils of babies. The dilation will last for about 6 to 10 hours. After the test, the baby will return to the nursery or be discharged home as intended by the Neonatology Division.

There is minimal risk associated with this investigation. The instrument is non-invasive and does not touch the eye. The babies will be swaddled and held by a nurse to prevent any contact with the machine. The eye drop to be used if needed for dilation has been used on babies at Harbor for about 30 years. It has been found to very safe. The fact that we will study only term (not premature babies) and will apply only two drops if needed should minimize any risk from the eye drop.

An ethical issue to consider is that while the study will provide important information that will undoubtedly help babies in the future, it will probably not benefit the baby being studied. However, if the baby has an undetected retinal or optic nerve problem, the study may reveal it.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term, gestational age of 38-42 weeks inclusive.
* Able to be transported to the Eye Clinic.
* No longer monitored. On no intravenous or other lines.

Exclusion Criteria:

* History of hyperglycemia in the infant (a blood sugar greater than 100mg%, per Laboratory Policy on Critical Values for infants less than 20 days old).
* Feeding intolerance.
* Green-tinged aspirates/emesis.
* Abdominal distention.
* History of genetic consult indicating any abnormality.
* Any known ocular disorder.

Ages: 38 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Specific eye measurements by SD-OCT, including retinal nerve fiber layer thickness per quadrant, foveal depth, optic cup area and depth, optic nerve/foveal distance and depth of various layers within the retina to determine neonatal baseline values. | 24 months
  A spreadsheet of the data collected from the study population will be created. The data will be derived from analysis of the images captured by the instrument. Software within the computer of the instrument will provide data from each image including measurements of retinal nerve fiber layer thickness in each quadrant, depth of the fovea, depth and area of the optic cup, distance from the optic nerve to the fovea, and depth of the various layers within the retina. These parameters will be calculated to establish normal values for the first time.

CONTACTS AND LOCATIONS:
Overall Officials: Sherwin J Isenberg, M.D., Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Los Angeles Biomedical Research Institute atHarbor-UCLA Medical Center, Torrance, California, United States